CLINICAL TRIAL: NCT05992493
Title: To Explore and Develop the Effective Human Milk Oligosaccharides and Microbiomes on Maternal and Infant Health and Neurodevelopment in Early Infancy
Brief Title: The Role of Human Milk Oligosaccharides and Microbiomes on Infantile Colic and Atopic Dermatitis in Term Infants
Status: Active, not recruiting | Type: Observational
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Principal Investigator, Yao-Jong Yang, professor, National Cheng-Kung University Hospital
Other Study IDs: A-BR-109-005
Record Dates: First submitted 2022-09-30; First posted 2023-08-15 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Infantile Colic; Breast Feeding; Atopic Dermatitis; Infant Formula
Keywords: Breast milk; microbiota; infant health; Human milk oligosaccharides; prebiotics
MeSH Terms: conditions — Colic; Breast Feeding; Dermatitis, Atopic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — infant fecal sample and mother breast-milk sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Breast-milk feeding: Exclusive breastfeeding for 4 months or more
- Control Formula milk feeding: Exclusive formula milk for 4 months or more
- HMO-Formula-milk feeding: Exclusive HMO-formula milk for 4 months or more

SUMMARY:
Background: Human milk oligosaccharides (HMO) and microbiota are both key factors for infants to shape the gut flora and develop the immune system. Breastfed infant is beneficial to prevent the occurrence of infantile colic (IC) and atopic dermatitis (AD), which may through shaping a healthy microbiota. However, the gut microbiota biomarkers representing IC and AD have not yet been discovered. In addition, the effectiveness of supplement of HMO in infant formula reduce the incidence of IC and AD in infants is still debate.

DETAILED DESCRIPTION:
Purpose: To investigate the preventive role of HMO-supplement formula on IC and AD in term infants in a clinical trial.

Method: The investigators will enroll three cohorts (exclusive breastfeeding, formula feeding, and HMO-supplement formula feeding infants) for research. The investigators collected samples of serial baby feces from subjects at 0, 1, 2, 4, 6, 12 months in this study. The fecal microbiota composition will be analyzed by detecting 16S-rRNA using next generation sequencing method. The demographic data and incidence of IC (0-5 months) and AD (0-12 months) was followed and recorded.

ELIGIBILITY:
Inclusion Criteria:

1. New born
2. Gestational age of >= 37 weeks
3. birth weight greater than 2500 gm

Exclusion Criteria:

1. Born with Perinatal insults
2. Mother with antimicrobial agents 1 month before delivery
3. Congenital abnormalities related to growth
4. Major disease admitted to Level II or NICU

Min Age: 1 Day | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The investigators collected exclusive, formula-fed and HMO-supplement formula-fed infants. Inclusion criteria were infants with a gestational age >= 37 weeks and a birth weight greater than 2500 gm. Exclusion criteria were infants born with perinatal injury, use of antibiotics prior to stool collection, growth-related congenital anomalies, and major illnesses requiring hospitalization.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-08-07 (Actual); Primary Completion 2025-08-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of IC and AD will be compared between three groups | The 1 months after birth follow-up
  According to the feeding method, singleton full-term infants will divide into three groups (n=300) including recorded demographic data. The diagnosis of IC and AD is based on Rome IV criteria and the Taiwan Academy of Pediatric Allergy, Asthma, and Immunology (TAPAAI) criteria, respectively. The incidence of IC and AD will be compared between the three groups.
Incidence of IC and AD will be compared between three groups | The 2 months after birth follow-up
  According to the feeding method, singleton full-term infants will divide into three groups (n=300) including recorded demographic data. The diagnosis of IC and AD is based on Rome IV criteria and the Taiwan Academy of Pediatric Allergy, Asthma, and Immunology (TAPAAI) criteria, respectively. The incidence of IC and AD will be compared between the three groups.
Incidence of IC and AD will be compared between three groups | The 4 months after birth follow-up
  According to the feeding method, singleton full-term infants will divide into three groups (n=300) including recorded demographic data. The diagnosis of IC and AD is based on Rome IV criteria and the Taiwan Academy of Pediatric Allergy, Asthma, and Immunology (TAPAAI) criteria, respectively. The incidence of IC and AD will be compared between the three groups.
Incidence of IC and AD will be compared between three groups | The 6 months after birth follow-up
  According to the feeding method, singleton full-term infants will divide into three groups (n=300) including recorded demographic data. The diagnosis of IC and AD is based on Rome IV criteria and the Taiwan Academy of Pediatric Allergy, Asthma, and Immunology (TAPAAI) criteria, respectively. The incidence of IC and AD will be compared between the three groups.
Incidence of IC and AD will be compared between three groups | The 12 months after birth follow-up
  According to the feeding method, singleton full-term infants will divide into three groups (n=300) including recorded demographic data. The diagnosis of IC and AD is based on Rome IV criteria and the Taiwan Academy of Pediatric Allergy, Asthma, and Immunology (TAPAAI) criteria, respectively. The incidence of IC and AD will be compared between the three groups.
Next-generation sequencing analysis-based differences on gut microbiota in infants between three groups | Infant stool samples will be collected at various time points from 0 to 1 year of age.
  Singleton full-term infants will divide into three groups (n=300) according to feeding method. The collected fecal samples will be analyze the composition of microbiota using NGS method. The differences of microbiota pattern will be identified.

SECONDARY OUTCOMES:
Infantile weight growth between different feeding pattern | The 1 months after birth follow-up
  Singleton full-term infants will divide into three groups (n=300) according to feeding method. The body weight growth (gm) will be recorded and compared between the three groups.
Infantile weight growth between different feeding pattern | The 2 months after birth follow-up
  Singleton full-term infants will divide into three groups (n=300) according to feeding method. The body weight growth (gm) will be recorded and compared between the three groups.
Infantile weight growth between different feeding pattern | The 4 months after birth follow-up
  Singleton full-term infants will divide into three groups (n=300) according to feeding method. The body weight growth (gm) will be recorded and compared between the three groups.
Infantile weight growth between different feeding pattern | The 6 months after birth follow-up
  Singleton full-term infants will divide into three groups (n=300) according to feeding method. The body weight growth (gm) will be recorded and compared between the three groups.
Infantile weight growth between different feeding pattern | The 12 months after birth follow-up
  Singleton full-term infants will divide into three groups (n=300) according to feeding method. The body weight growth (gm) will be recorded and compared between three groups.
Infantile height growth between different feeding pattern | The 1 months after birth follow-up
  Singleton full-term infants will divide into three groups (n=300) according to feeding method. The body height growth (cm) will be recorded and compared between the three groups.
Infantile height growth between different feeding pattern | The 2 months after birth follow-up
  Singleton full-term infants will divide into three groups (n=300) according to feeding method. The body height growth (cm) will be recorded and compared between the three groups.
Infantile height growth between different feeding pattern | The 4 months after birth follow-up
  Singleton full-term infants will divide into three groups (n=300) according to feeding method. The body height growth (cm) will be recorded and compared between the three groups.
Infantile height growth between different feeding pattern | The 6 months after birth follow-up
  Singleton full-term infants will divide into three groups (n=300) according to feeding method. The body height growth (cm) will be recorded and compared between the three groups.
Infantile height growth between different feeding pattern | The 12 months after birth follow-up
  Singleton full-term infants will divide into three groups (n=300) according to feeding method. The body height growth (cm) will be recorded and compared between the three groups.

CONTACTS AND LOCATIONS:
Locations (1):
- National Cheng Kung University & Hospital, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Zivkovic AM, German JB, Lebrilla CB, Mills DA. Human milk glycobiome and its impact on the infant gastrointestinal microbiota. Proc Natl Acad Sci U S A. 2011 Mar 15;108 Suppl 1(Suppl 1):4653-8. doi: 10.1073/pnas.1000083107. Epub 2010 Aug 2. PMID 20679197
- [Background] Le Doare K, Holder B, Bassett A, Pannaraj PS. Mother's Milk: A Purposeful Contribution to the Development of the Infant Microbiota and Immunity. Front Immunol. 2018 Feb 28;9:361. doi: 10.3389/fimmu.2018.00361. eCollection 2018. PMID 29599768
- [Background] Ward RE, Ninonuevo M, Mills DA, Lebrilla CB, German JB. In vitro fermentation of breast milk oligosaccharides by Bifidobacterium infantis and Lactobacillus gasseri. Appl Environ Microbiol. 2006 Jun;72(6):4497-9. doi: 10.1128/AEM.02515-05. PMID 16751577